CLINICAL TRIAL: NCT04164654
Title: Using a Mobile App to Address Student Loneliness Among College Students: A Randomized Controlled Trial
Brief Title: A Mobile App to Address Student Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: HopeLab Foundation (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06072019.014; R34DA041637 (NIH)
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Immediate Access to the Nod app (Experimental): The experimental group will have immediate access to all content in the Nod app and will be free to engage with it as much or as little as they like for four weeks. They will retain access to the Nod app for an additional four weeks.
  Interventions: Behavioral: Loneliness Intervention
- Waitlist Control-Delayed Access to the Nod app (Other): The waitlist control group will have full access to the Nod app approximately four weeks after the experimental group gains access.
  Interventions: Behavioral: Loneliness Intervention

INTERVENTIONS:
Behavioral: Loneliness Intervention — 28 days of engagement with the Nod app, which consists of interactive exercises drawn from cognitive behavioral therapy (e.g behavioral activation and cognitive reframing exercises), positive psychology (e.g. acts of kindness), and mindful self-compassion programs (e.g. loving-kindness meditations)
  Other Names: A mobile app called Nod

SUMMARY:
The purpose of this trial is to assess the effects of a positive psychology and CBT-based skills intervention-delivered through a mobile app called Nod-on loneliness and other mental health and institutional satisfaction outcomes. The primary outcome is self-reported loneliness at 2 and 4-weeks post baseline.

DETAILED DESCRIPTION:
This study is a pilot eight-week randomized controlled intervention. It employs a "waitlist" control strategy for the first 4 weeks of the study (considered to be the active study period).

Randomization will be to one of two conditions:

1. Experimental group: Immediate access to the Nod app
2. Waitlist control group: Participants will be granted access to the app four weeks after the experimental group

Assessments will occur at baseline, 2, 4, and 8 weeks follow up. Assessments will include measures of loneliness, and other mental health and institutional satisfaction measures listed in the secondary outcome measures section.

ELIGIBILITY:
Inclusion Criteria:

* Incoming college first years
* Live away from home without parents/guardians upon beginning college
* Read English
* Between 18 and 25 years of age
* Own a smartphone

Exclusion Criteria:

* Do not read English
* Under 18 years of age
* Over 25 years of age
* Do not own a smartphone

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Condition differences in self-reported loneliness | 2-weeks post baseline
  Total score on the UCLA-8. Scores range from 8-32, higher scores indicate worse depression.
Condition differences in self-reported loneliness | 4-weeks post baseline
  Total score on the UCLA-8. Scores range from 8-32, higher scores indicate worse depression.

SECONDARY OUTCOMES:
Depressive symptoms | 2 and 4 weeks post baseline
  Total score on the Patient Health Questionnaire 9-item scale. Scores range from 0-27, higher scores indicate worse depression.
Anxiety | 2 and 4 weeks post baseline
  Total score on the Generalized Anxiety Disorder 7-item scale. Scores range from 0-21, higher scores indicate worse anxiety.
Social Anxiety | 2 and 4 weeks post baseline
  Total score on the Mini Social Phobia Inventory. Scores range from 0-12, higher scores indicate worse social anxiety.
Self-reported intention to remain enrolled at the University of Oregon in the next academic year | 2 and 4 weeks post baseline
  Self-reported intention to remain enrolled at the University of Oregon in the next academic year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruehlman-Senecal E, Hook CJ, Pfeifer JH, FitzGerald C, Davis B, Delucchi KL, Haritatos J, Ramo DE. Smartphone App to Address Loneliness Among College Students: Pilot Randomized Controlled Trial. JMIR Ment Health. 2020 Oct 20;7(10):e21496. doi: 10.2196/21496. PMID 33079071